CLINICAL TRIAL: NCT00292526
Title: Prevention of Chemotherapy-induced Cardiotoxicity in High-risk Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: IEO S67/500
Record Dates: First submitted 2006-02-15; First posted 2006-02-16 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Cardiotoxicity; Chemotherapeutic Toxicity
Keywords: Chemotherapy induced cardiotoxicity; Troponin; Heart failure
MeSH Terms: conditions — Cardiotoxicity; Heart Failure | interventions — Enalapril

ARMS (1):
- enalapril arm (Experimental): treatment with enalapril
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Enalapril — enalapril orally administered

SUMMARY:
In cancer patients, the increase of troponin I soon after chemotherapy is a strong predictor of left ventricular dysfunction and poor cardiologic outcome. This information provides a rationale for the development of prophylactic strategies directed against chemotherapy-induced cardiotoxicity (CTIC). Activation of the renin-angiotensin system has been proved to be involved in the development and progression of cardiac dysfunction in several clinical settings, and has been suggested to have a role in the occurrence of CTIC. We investigated the role of treatment with ACE-inhibitors in the prevention of CTIC in high-risk cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients undergoing high-dose chemotherapy showing early release of Troponin I

Exclusion Criteria:

* Contraindication to ACE-inhibitors
* On-going therapy with beta-blockers, ACE-inhibitors, angiotensin-receptors blockers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2000-11 (Actual); Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Incidence of chemotherapy-induced cardiotoxicity | 12 month period

SECONDARY OUTCOMES:
Major adverse cardiac events, including death. | 12 month period

CONTACTS AND LOCATIONS:
Overall Officials: Carlo M Cipolla, MD, Study Director — European Institute of Oncology; Daniela Cardinale, MD, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cardinale D, Sandri MT, Colombo A, Colombo N, Boeri M, Lamantia G, Civelli M, Peccatori F, Martinelli G, Fiorentini C, Cipolla CM. Prognostic value of troponin I in cardiac risk stratification of cancer patients undergoing high-dose chemotherapy. Circulation. 2004 Jun 8;109(22):2749-54. doi: 10.1161/01.CIR.0000130926.51766.CC. Epub 2004 May 17. PMID 15148277
- [Background] Cardinale D, Sandri MT, Martinoni A, Tricca A, Civelli M, Lamantia G, Cinieri S, Martinelli G, Cipolla CM, Fiorentini C. Left ventricular dysfunction predicted by early troponin I release after high-dose chemotherapy. J Am Coll Cardiol. 2000 Aug;36(2):517-22. doi: 10.1016/s0735-1097(00)00748-8. PMID 10933366